CLINICAL TRIAL: NCT03460041
Title: Caudal Dexmetedomedine Versus Magnesium in Orthopedic Pediatric Surgeries
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hagar hassanein refaee (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Hagar hassanein refaee, Assistant lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: N-59-2017
Record Dates: First submitted 2018-02-26; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Pain in Pediatric Patients
MeSH Terms: interventions — Magnesium Sulfate; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator)
  Interventions: Drug: Bupivacaine
- Magnesium (Active Comparator)
  Interventions: Drug: Magnesium Sulfate
- Dexmetedomedine (Active Comparator)
  Interventions: Drug: Dexmetedomedine

INTERVENTIONS:
Drug: Magnesium Sulfate — caudal magnesium sulphate added to bupivacaine for pain management
  Arms: Magnesium
Drug: Dexmetedomedine — Caudal dexmetedomedine added to bupivacaine for pain management
  Arms: Dexmetedomedine
Drug: Bupivacaine — Caudal bupivacaine for pain management
  Arms: Control

SUMMARY:
This study will be performed in Abo Elreesh Pediatric Hospital / Cairo University after obtaining approval by the University Ethics Committee, and a written informed consent from the parents or guardians.

Thirty six patients will be randomly assigned using an online randomization program (http://www.randomizer.org) and the sealed envelope method into three groups: Group D (n=12): Dexmetedomidine group. 0.5 ml of dexmetedomidine (2 μg/kg) added to bupivacaine, Group M (n=12) : Magnesium group.0.5 ml of magnesium sulphate (50 mg) added to bupivacaine, Group C (n=12) :Control group.bupivacaine 0.25% diluted in normal saline with total volume of 1 ml/kg.

DETAILED DESCRIPTION:
History regarding previous anesthesia, surgery, any significant medical illness, medications and allergy will be taken for all children who will be enrolled in the study. Complete physical examination and airway assessment will be done. Hemoglobin percentage, blood sugar and coagulation profile will be investigated preoperatively Sedation will be done by giving midazolam (0.2 mg/kg IM).On arrival to the operating room all patients will be monitored by 5 leads electrocardiography (ECG), automated non-invasive blood pressure monitoring (NIBP), and pulse oximetery.

Inhalational induction of anesthesia will be achieved by 8% sevoflurane in 100% oxygen and an appropriate-sized cannula will be inserted. Endotracheal intubation will be performed after which sevoflurane concentration will be reduced to 3%. After hemodynamic stabilization, caudal block will be performed by using beveled needle 18-23 G in the lateral decubitus position by using the loss of resistance technique. The study solutions will be injected caudally slowly with repetitive intermittent aspiration by an anesthesiologist blinded to the test drugs. The inhaled concentration of sevoflurane will be adjusted to achieve hemodynamic changes less than 30% of the preoperative values

Recorded Parameters for the study:

Intraoperative hemodynamic: heart rates (beats/minutes), mean arterial blood pressure (mmHg) after stabilization, before skin incision and every 15 minutes till the end of surgery.

Sedation score: Sedation will be monitored after PACU arrival using Ramsay score with its 0-6 score range.

Pain score (FLACC score) with its 0-10 score range, each patient pain intensity will be assessed at the end of surgery and 12 hours postoperatively.

Time of rescue analgesia (from the time of caudal injection to the time at which FLACC score 4 or more) will be recorded.

Complication secondary to test drugs in the form of toxicity like postoperative nausea and vomiting, respiratory depression, hematoma, bradycardia (HR <80 BPM) and hypotension (SBP <70 mmhg+ age in years * 2) and complication secondary to caudal block; infection, hematoma and pain at the site of injection will be recorded.

Total doses of rescue drugs will be calculated for each group.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 - 7 years old.
* American Society of Anesthesiologist (ASA) physical status class I- II.
* Patients scheduled for infra-umbilical orthopedic surgeries.

Exclusion Criteria:

* Patients with known allergy to the study drugs
* Suspected coagulopathy.
* Infection at the site of caudal block.
* History of developmental delay or neuromuscular disorders.
* Skeletal deformities.
* Patients on magnesium therapy

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-03-15 (Estimated); Study Completion 2018-03-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 12 hours
  Comparing duration of analgesia between caudal magnesium and caudal dexmetedomedine using flacc score

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University faculty, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No